CLINICAL TRIAL: NCT02383927
Title: An Open Label Phase II Study of Tipifarnib in Advanced Non-Hematological Malignancies With HRAS Mutations
Brief Title: Phase II Study of Tipifarnib in Squamous Head and Neck Cancer With HRAS Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KO-TIP-001
Record Dates: First submitted 2015-02-20; First posted 2015-03-10 (Estimated); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Thyroid Cancer; Squamous Cell Carcinoma Head and Neck Cancer (HNSCC); HRAS Mutant Tumor; Other Squamous Cell Carcinoma (SCC) With HRAS Mutant Tumor
MeSH Terms: conditions — Thyroid Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Thyroid Cancer
  Interventions: Drug: Tipifarnib
- Cohort 2 (Experimental): Squamous Head and Neck Cancer
  Interventions: Drug: Tipifarnib

INTERVENTIONS:
Drug: Tipifarnib — FTase inhibitor
  Other Names: Zarnestra

SUMMARY:
Phase II study to investigate the antitumor activity in terms of objective response rate (ORR) of tipifarnib in subjects with advanced tumors that carry HRAS mutations and for whom there is no standard curative therapy available.

DETAILED DESCRIPTION:
This Phase II study will investigate the antitumor activity in terms of ORR of tipifarnib in subjects with locally advanced, unresectable or metastatic, relapsed and/or refractory tumors that carry HRAS mutations and for whom there is no curative therapy available. Subjects with information available on tumor HRAS status previously generated are eligible. All subjects must consent to provide at least 10 tumor slides from a prior diagnostic biopsy for a retrospective testing of HRAS gene status at a central facility.

Subjects will be enrolled into three nonrandomized cohorts:

* Cohort 1: Malignant thyroid tumors with HRAS mutations.
* Cohort 2: Squamous Cell Carcinoma Head and Neck Cancer with HRAS mutations.
* Cohort 3: Squamous Cell Carcinoma (SCC) with HRAS mutations other than HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed diagnosis of thyroid cancer (cohort 1) or Squamous Cell Carcinoma head and neck cancer (cohort 2) or Squamous Cell Carcinoma other than HNSCC (cohort 3) for which there is no curative therapy available.
* tumor that carries a missense HRAS mutation ith a variant allele frequency (VAF) > 20%.
* Subject consents to provide at least 10 unstained tumor slides for retrospective testing of HRAS gene tumor status
* Subject has measurable disease according to RECIST v1.1 and has relapsed or is refractory to prior therapy.
* At least 2 weeks since the last systemic therapy or radiotherapy regimen prior to enrolment
* ECOG PS 0 or 1
* Acceptable liver function
* Acceptable renal function
* Acceptable hematologic status • Serum albumin ≥ 3.5 g/dL. Subjects with tumors potentially highly sensitive to tipifarnib (HRAS mutant VAF ≥ 35%) may be enrolled despite a serum albumin < 3.5 g/dL.

Exclusion Criteria:

* Prior treatment with an FTase inhibitor
* History of relevant coronary heart disease or myocardial infarction within last 3 years, NYHA Grade III or greater congestive heart failure, cerebro-vascular attack within the prior year, or serious cardiac arrhythmia requiring medication except atrial fibrillation.
* Known uncontrolled brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 4 weeks prior to Cycle 1 Day 1). Controlled brain metastases that require continuous high dose corticosteroid use within 4 weeks of Day 1.
* Non-tolerable > Grade 2 neuropathy or evidence of unstable neurological symptoms within 4 weeks first dose
* Major surgery, other than diagnostic surgery, within 4 weeks prior to first dose, without complete recovery.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy. Known infection with HIV, or an active infection with hepatitis B or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-05-13; Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (9):
  - University of California, Los Angeles, Los Angeles, California
  - Wihship Cancer Institute of Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (3):
  - University Hospital Antwerp, Antwerp
  - Cliniques universitaires Saint-Luc, Brussels
  - CHU, Yvoir
- France (4):
  - Insitut Bergonie, Bordeaux
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institute Gustave Roussy (IGR), Paris
- University Hospital Wuerazburg, Würzburg, Germany
- Attikon University Hospital, Attiki, Greece
- Instituto Nazionale Tumori, Milan, Italy
- University Medical Center, Groningen, Netherlands
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (11):
  - Hospital Vall d' Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - START, Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complejo Hospitalario de Navarro, Navarro
  - Hospital Universitario Virgen de la Rocio, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (2):
  - Royal Marsden, London, England
  - University College Hospital, London, England

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ho AL, Brana I, Haddad R, Bauman J, Bible K, Oosting S, Wong DJ, Ahn MJ, Boni V, Even C, Fayette J, Flor MJ, Harrington K, Kim SB, Licitra L, Nixon I, Saba NF, Hackenberg S, Specenier P, Worden F, Balsara B, Leoni M, Martell B, Scholz C, Gualberto A. Tipifarnib in Head and Neck Squamous Cell Carcinoma With HRAS Mutations. J Clin Oncol. 2021 Jun 10;39(17):1856-1864. doi: 10.1200/JCO.20.02903. Epub 2021 Mar 22. PMID 33750196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with thyroid cancer with Harvey Rat sarcoma virus (HRAS) mutations were enrolled in Cohort 1; subjects with any solid tumour with HRAS mutation were enrolled in Stage 1 of Cohort 2; subjects with head and neck squamous cell carcinoma (HNSCC) with HRAS mutations were enrolled in Stage 2 of Cohort 2; subjects with any squamous cell carcinoma (SCC) (excluding HNSCC) with HRAS mutation were enrolled in Cohort 3.
Pre-assignment Details: Only consented subjects who met all the eligibility criteria were enrolled in the study. All screening evaluations were to be completed within 4 weeks (28 days) of Cycle 1 Day 1.
Groups:
- Cohort 1: Subjects with thyroid cancer with HRAS mutations.
  Subjects received tipifarnib as monotherapy orally twice daily (BID) on Days 1-7 and 15-21 of each 28-day treatment cycle.
  In the absence of unacceptable tipifarnib-related emergent toxicity or disease progression, subjects could receive treatment with tipifarnib for up to 12 months at the discretion of the Investigator. Treatment beyond 12 months may have continued upon agreement of the Investigator and the Sponsor.
- Cohort 2/Stage 1: Subjects with any solid tumour with HRAS mutation.
  Subjects received tipifarnib as monotherapy orally BID on Days 1-7 and 15-21 of each 28-day treatment cycle.
  In the absence of unacceptable tipifarnib-related emergent toxicity or disease progression, subjects could receive treatment with tipifarnib for up to 12 months at the discretion of the Investigator. Treatment beyond 12 months may have continued upon agreement of the Investigator and the Sponsor.
- Cohort 2/Stage 2: Subjects with HNSCC with HRAS mutations.
  Subjects received tipifarnib as monotherapy orally BID on Days 1-7 and 15-21 of each 28-day treatment cycle.
  In the absence of unacceptable tipifarnib-related emergent toxicity or disease progression, subjects could receive treatment with tipifarnib for up to 12 months at the discretion of the Investigator. Treatment beyond 12 months may have continued upon agreement of the Investigator and the Sponsor.
- Cohort 3: Subjects with any SCC (excluding HNSCC) with HRAS mutation.
  Subjects received tipifarnib as monotherapy orally BID on Days 1-7 and 15-21 of each 28-day treatment cycle.
  In the absence of unacceptable tipifarnib-related emergent toxicity or disease progression, subjects could receive treatment with tipifarnib for up to 12 months at the discretion of the Investigator. Treatment beyond 12 months may have continued upon agreement of the Investigator and the Sponsor.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3
Started | 13 | 10 | 30 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 13 | 10 | 30 | 10
Not completed — Disease Progression | 8 | 8 | 15 | 4
Not completed — Physician Decision | 0 | 0 | 2 | 0
Not completed — Termination by Symptomatic Deterioration | 0 | 0 | 6 | 0
Not completed — Adverse Event | 4 | 1 | 3 | 5
Not completed — Miscellaneous | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: The All Subjects as Treated (ASaT) Population consists of all enrolled subjects who received at least 1 dose of tipifarnib.
Groups:
- Cohort 1: Subjects with thyroid cancer with HRAS mutations.
  Subjects received tipifarnib as monotherapy orally BID on Days 1-7 and 15-21 of each 28-day treatment cycle.
  In the absence of unacceptable tipifarnib-related emergent toxicity or disease progression, subjects could receive treatment with tipifarnib for up to 12 months at the discretion of the Investigator. Treatment beyond 12 months may have continued upon agreement of the Investigator and the Sponsor.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3 | Total
Number analyzed (Participants) | 13 | 10 | 30 | 10 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (7.4) | 59.1 (16.9) | 61.0 (14.4) | 67.0 (11.7) | 65.32 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 8 | 5 | 19
  Male | 9 | 8 | 22 | 5 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 3
  Not Hispanic or Latino | 12 | 10 | 28 | 10 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 7 | 24 | 10 | 48
  Black or African American | 2 | 1 | 1 | 0 | 4
  Asian | 2 | 1 | 4 | 0 | 7
  Other | 2 | 1 | 1 | 0 | 4
Eastern Cooperative Oncology Group (ECOG) performance score [Count of Participants; unit: Participants] — Performance Score:
  * 0: Fully active, able to carry on all predisease performance without restriction.
  * 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    Performance score 0 | 7 | 3 | 3 | 1 | 14
    Performance score 1 | 6 | 7 | 27 | 9 | 49
Type of tumour [Count of Participants; unit: Participants]
  Thyroid | 13 | 0 | 0 | 0 | 13
  Head and neck | 0 | 0 | 30 | 0 | 30
  Salivary | 0 | 7 | 0 | 0 | 7
  Skin | 0 | 0 | 0 | 4 | 4
  Other | 0 | 3 | 0 | 6 | 9
Stage of cancer [Count of Participants; unit: Participants] — Cancer stages:
  * Stage I: early stage; a small invasive mass or tumor, no spread to lymph nodes or other issues.
  * Stage II: localized; cancer has started to affect nearby tissues, mass may have grown in size, spread to lymph nodes near the mass.
  * Stage III: region spread; cancer affects more surrounding tissue, mass may have grown in size, spread to distant lymph nodes.
  * Stage IV: distant spread; cancer has spread to other tissues or organs beyond the region where it originated, considered "metastatic".
  Participants
    Stage I | 0 | 0 | 0 | 1 | 1
    Stage II | 0 | 0 | 2 | 0 | 2
    Stage III | 1 | 1 | 2 | 0 | 4
    Stage IV | 12 | 9 | 26 | 9 | 56

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Activity by Objective Response Rate (ORR)
Description: The ORR of tipifarnib was response assessments according to RECIST 1.1. The estimate of the ORR was calculated based on the maximum likelihood estimator (i.e., crude percentage of subjects whose best overall response was complete response [CR] or partial response [PR]). The estimate of the ORR was accompanied by 2-sided 95% confidence interval (CI). The 95% CI was estimated using the Wilson score test-based method.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (< 10 mm short axis).
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: Up to approximately 3 years
Population: The Full Analysis Set (FAS) Population excluding subjects for the following reasons: no baseline data; failure to receive at least 1 dose of tipifarnib; no post-baseline endpoint data subsequent to at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3
Number analyzed (Participants) | 11 | 8 | 23 | 7
percentage of participants | 0.0 [0.0 to 25.9] | 0.0 [0.0 to 32.4] | 43.5 [25.6 to 63.2] | 28.6 [8.2 to 64.1]

2. Secondary Outcome: Number of Subjects That Experienced One or More Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs that started on or after the first dose of study drug and within 30 days of the last administration of study drug or immediately before the initiation of any other anticancer therapy. The Investigator was required to grade the severity/ intensity of each AE according to NCI-CTCAE version 4.03. If a severity/intensity of Grade 4 (life-threatening) or 5 (death) was applied to an AE, then the Investigator also reported the event as a serious AE.
Time Frame: Up to approximately 3 years
Population: The ASaT Population consists of all enrolled subjects who received at least 1 dose of tipifarnib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3
Number analyzed (Participants) | 13 | 10 | 30 | 10
Participants
  TEAEs | 13 | 10 | 30 | 10
  Serious TEAEs | 6 | 5 | 20 | 9

3. Other Pre Specified Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from first dose (Cycle 1 Day 1) to either first observation of progressive disease (PD) or occurrence of death due to any cause within 126 days (approximately 2 time-intervals for tumour assessments) of either first administration of tipifarnib or the last tumour assessment. Observation of PD could have been by either documented radiographic progression (i.e., scan results) or documentation of symptomatic or clinical progression agreed upon and documented by investigators. In subjects without a progression date or with a death date more than 126 days after the first administration of study drugs or the last tumour assessment, the PFS time should have been censored on the date of last tumour assessment or date of first administration of study tipifarnib.
Time Frame: Up to approximately 3 years
Population: The FAS Population excluding subjects for the following reasons: no baseline data; failure to receive at least 1 dose of tipifarnib; no post-baseline endpoint data subsequent to at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3
Number analyzed (Participants) | 11 | 8 | 23 | 7
months | 4.6 [3.1 to 8.4] | 6.4 [1.8 to 10.3] | 5.5 [3.6 to 9.2] | 8.0 [3.7 to 9.3]

4. Other Pre Specified Outcome: Duration of Response (DOR)
Description: DOR was the number of months from start date of PR or CR (whichever response was achieved first) to the first date that PD was documented (in subjects with an objective response). PD was determined by the Investigator using RECIST 1.1. The DOR was right-censored at the date for subjects who achieved CR or PR and met one of the following conditions: 1) when non-protocol anticancer treatment started before documentation of PD, 2) when death prior to documented PD or documented PD after more than 1 missed disease assessment visit, or 3) when alive and did not have documentation of PD before a data analysis cut-off date (therefore, analysis cut-off date was used as the censoring date). Median and 95% CI were calculated via Kaplan-Meier analysis.
Time Frame: Up to approximately 3 years
Population: The Per Protocol (PP) Population was a subset of the FAS population that excluded subjects due to major deviations from the protocol that may have substantially affected the results of the primary analysis. Only participants participants with response data were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 10 | 2
months |  |  | 6.2 [3.8 to 14.7] | NA [7.5 to NA] — Median and upper 95% CI were not reached as there were too few participants with events that impacted the estimate of DOR function.

5. Other Pre Specified Outcome: Overall Survival (OS)
Description: An analysis of OS was conducted to estimate median OS time and corresponding 95% CI. OS was defined as the time from first dose (Cycle 1 Day 1) to the occurrence of death due to any cause. In subjects without a death date, the OS was censored on 1) the last date of survival status if alive, 2) a data analysis cut-off date for subjects with no survival status documentation, or 3) the date a subject withdrew consent or was lost to follow-up if there was no additional information. Median and 95% CI were calculated via Kaplan-Meier analysis.
Time Frame: Up to approximately 4 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3
Number analyzed (Participants) | 11 | 8 | 23 | 7
months | 36.7 [8.7 to NA] — Upper 95% CI was not reached as there were too few participants with events that impacted the estimate of OS function. | 13.8 [5.3 to 29.9] | 10.8 [7.0 to 14.0] | 10.4 [6.2 to 16.1]

6. Other Pre Specified Outcome: Antitumor Activity - Best Overall Response (BOR)
Description: BOR according to RECIST 1.1.
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: Up to approximately 3 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3
Number analyzed (Participants) | 11 | 8 | 23 | 7
Participants
  CR | 0 | 0 | 0 | 0
  PR | 0 | 0 | 10 | 2
  SD | 9 | 6 | 11 | 4
  PD | 2 | 2 | 2 | 1
  Not evaluable | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: up to approximately 4 years; serious and other AEs: up to approximately 3 years
Arm/Group | Cohort 1 | Cohort 2/Stage 1 | Cohort 2/Stage 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 6/13 | 9/10 | 24/30 | 9/10
Serious Adverse Events (participants affected / at risk) | 6/13 | 5/10 | 20/30 | 9/10
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10 | 29/30 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=13) | Cohort 2/Stage 1 (N=10) | Cohort 2/Stage 2 (N=30) | Cohort 3 (N=10)
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 2
Discomfort (General disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=13) | Cohort 2/Stage 1 (N=10) | Cohort 2/Stage 2 (N=30) | Cohort 3 (N=10)
Hypertension (Vascular disorders) | 2 | 2 | 1 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 10 | 4 | 15 | 5
Asthenia (General disorders) | 1 | 1 | 6 | 2
Pyrexia (General disorders) | 1 | 3 | 4 | 0
Oedema peripheral (General disorders) | 1 | 2 | 4 | 0
Pain (General disorders) | 0 | 1 | 5 | 1
Chills (General disorders) | 1 | 1 | 1 | 0
Face oedema (General disorders) | 1 | 0 | 2 | 0
Malaise (General disorders) | 0 | 1 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 2 | 2
Insomnia (Psychiatric disorders) | 3 | 2 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 1
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 4 | 7 | 5
Weight decreased (Investigations) | 3 | 2 | 7 | 0
Blood bilirubin increased (Investigations) | 2 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 2 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0 | 0 | 0
Blood urea increased (Investigations) | 2 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 1 | 0
Protein urine present (Investigations) | 2 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0
Blood calcitonin increased (Investigations) | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 3 | 2 | 3 | 1
Platelet count decreased (Investigations) | 4 | 5 | 4 | 2
White blood cell count decreased (Investigations) | 3 | 3 | 5 | 3
Neutrophil count decreased (Investigations) | 0 | 3 | 5 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 2 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 9 | 5 | 19 | 6
Neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 3 | 0
Lymphocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 6 | 1
Headache (Nervous system disorders) | 2 | 1 | 2 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 2 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 2 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0 | 1
Asthenopia (Eye disorders) | 0 | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Ocular hypertension (Eye disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 5 | 16 | 2
Vomiting (Gastrointestinal disorders) | 4 | 2 | 14 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 10 | 3
Constipation (Gastrointestinal disorders) | 5 | 5 | 8 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 5 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 6 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are agreements in place between clinical trial sites and the Sponsor (or its agents) that govern discussion or publication of trial results by the sites or their employees after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02383927/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT02383927/SAP_001.pdf